CLINICAL TRIAL: NCT00172666
Title: Investigating Genetic Polymorphism of Decoy Receptor 3 (DcR3) Gene in Rheumatoid Arthritis and Systemic Lupus Erythematosus
Brief Title: Decoy Receptor 3 (DcR3) Polymorphisms in Rheumatoid Arthritis (RA) and Systemic Lupus Erythematosus (SLE)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701218; NSC 94-2320-B-002-085
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2006-03-30 (Estimated); Status verified 2004-12

CONDITIONS: Rheumatoid Arthritis; Systemic Lupus Erythematosus
Keywords: SLE; healthy subjects
MeSH Terms: conditions — Arthritis, Rheumatoid; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Although SLE and RA are correlated with genetic predisposing factors such as human leukocyte antigen (HLA) class II, both diseases and other genetic factors might have contributed to the development of dysregulated lymphocyte activation and autoimmunity.

Decoy receptor 3 (DcR3)/TR6 is a secreted protein belonging to the tumor necrosis factor (TNF) receptor family. It binds to Fas ligand (FasL), LIGHT, and TL1A that are all TNF family members. It was noted that soluble or solid phase DcR3-Fc co-stimulated proliferation, lymphokine production and cytotoxicity of mouse and human T cells upon T-cell receptor (TCR) ligation. Recently, the investigators found that the serum level of soluble DcR3 was higher in SLE patients than in healthy control subjects (unpublished data). Taken together, the investigators propose that in autoimmune diseases, such as RA and SLE, activated T cells secrete more DcR3 than non-autoimmune controls, which may, in turn, costimulate T cells further and cause dysregulated lymphocyte activation. With the aim to establish the possible correlation between DcR3 genetic polymorphisms, DcR3 expressions, and autoimmune phenotypes, the investigators offer this proposal. They plan to investigate the single nucleotide polymorphisms (SNPs) in the DcR3 gene. The genetic polymorphisms on the DcR3/TR6 gene and circulating DcR3 level will be compared between RA, SLE and non-autoimmune control subjects.

DETAILED DESCRIPTION:
Abnormal immune responses permit sustained production of pathogenic subsets of autoantibodies such as anti-DNA, and anti-RNP, anti-RBC, anti-platelet. T cell help is critical to development of full-blown disease; CD4+, CD8+, CD4-, CD8- lymphocytes all help autoantibody production in SLE. There are multiple abnormalities that permit hyper-activated self-reactive B and T cells to dominate the immune repertoire. Defects in cell activation, tolerance, apoptosis, idiotypic networks, immune complex clearance and generation of regulatory cells are all accounted for. SLE may involve only one organ system at disease onset or may be multi-systemic. Rheumatoid inflammation reflexes cause persistent stimulation of T cells by synovial-derived antigens that cross-react with determinants introduced during antecedent exposure to foreign antigens or infectious agents.

Decoy receptor 3 (DCR3/TR6) is a soluble, secreted factor that lacks a trans-membrane domain. It belongs to the TNFR family and is capable of binding to TNF family members FasL, LIGHT and TL1A. DcR3/TR6 mRNA is expressed at high levels in lymph nodes, the spleen and activated T cells. DcR3/TR6 binds to FasL and inhibits the Fas-FasL interaction and FasL-mediated apoptosis of lymphocytes and several tumor cell lines. LIGHT is highly expressed on surface of activated T lymphocytes and macrophages, CD8+ tumor-infiltrating lymphocyte, granulocytes and monocytes but not in the thymus and several human tumor cell lines. LIGHT protein triggers apoptosis of several tumor cells expressing both lymphotoxin β receptor (LTβR) and TR2. It was postulated that DcR3/TR6 modulated LIGHT-triggered costimulation via TR2 in T cells. Human PBMCs secrete DcR3/TR6 after PHA or anti-CD3. The leukocyte aggregation in mixed lymphocyte reaction was inhibited by adding soluble form DcR3. On the other hand, it was shown that DcR3/TR6, TR2, LIGHT displayed complexity in their interaction. The DcR3/TR6 expressed in solid phase actually transduced reverse, costimulatory signals into the activated T cells. Soluble DcR3-Fc or solid-phase DcR3-Fc was found to costimulate proliferation, lymphokine production and cytotoxicity of murine and human T cells in the presence of suboptimal TCR ligation. Furthermore, cross linking Th1 and Th2 cells with solid-phase DcR3-Fc along with suboptimal concentration of anti-CD3 enhanced proliferation of both Th1 and Th2 cells, and augmented Th1 but not Th2 cytokine production. These strongly suggest that DcR3/TR6 delivers costimulation through its ligand(s) on T cells, at least part of the costimulation is transduced via LIGHT. Recently, we found that soluble DcR3/TR6 level in circulating plasma in SLE patients was significantly higher than that of non-autoimmune control subjects. Plate-bound form DcR3 enhanced proliferation of T cells under suboptimal anti-CD3 stimulation in both normal and SLE patients. Addition of soluble DcR3-Fc reduced activation-induced cell death in T cells subjected to anti-CD3 re-stimulation (unpublished data). Taken together, it raises the possibility that genetic polymorphism in DcR3/TR6 locus might influence the expression level or function of DcR3, which in turn is implicated in dysregulated lymphocyte activation and autoimmunity. With the aim to establish the possible correlation between DcR3 genetic polymorphism, DcR3 expression, and autoimmune phenotypes, we give this proposal. We plan to investigate the single nucleotide polymorphisms (SNPs) in DcR3 gene. The genetic polymorphisms on DcR3/TR6 gene and circulating DcR3 level will be compared between RA, SLE and non-autoimmune control subjects.

The specific aims of this project are the following:

1. To study the allelic distribution of DcR3 genetic polymorphisms among the population in Taiwan.
2. To investigate if there is any DcR3 allele correlate to serum level of DcR3.
3. To investigate if the genetic polymorphism on DcR3 gene be associated with autoimmune diseases RA and SLE.

ELIGIBILITY:
Inclusion Criteria:

* SLE, RA, or healthy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2005-08; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Yi Hu, PhD, Principal Investigator — Department of Clinical Laboratory Sciences and Medical Biotechnology
Locations (1):
- Chung-Yi Hu, Taipei, Taiwan